CLINICAL TRIAL: NCT01034631
Title: Phase I/II Study of BNC105P in Combination With Everolimus or Following Everolimus For Progressive Metastatic Clear Cell Renal Cell Carcinoma Following Prior Tyrosine Kinase Inhibitors
Brief Title: BNC105P in Combination With Everolimus/Following Everolimus For Progressive Metastatic Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Bionomics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOG GU09-145
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2017-04

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic Kidney Cancer; BNC105P
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus; BNC 105P

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Arm A: Everolimus + BNC105P (Active Comparator): Combination Arm A: Everolimus 10 mg, BNC105P MTD (from Phase 1 study) 21 day cycle
  Interventions: Drug: Everolimus; Drug: BNC105P
- Sequential Arm B:Everolimus followed by BNC105P Monotherapy (Active Comparator): Sequential Arm B: Everolimus 10 mg, 21 day cycle
  Patients to receive BNC105P monotherapy at 16 mg/m2 following progression or intolerable toxicity on everolimus therapy.
  Interventions: Drug: Everolimus; Drug: BNC105P

INTERVENTIONS:
Drug: Everolimus — Everolimus 10 mg. Taken orally, every evening, 1 hr before or 2 hrs after meals
Drug: BNC105P — BNC105P, up to 16 mg/m^2

SUMMARY:
The purpose of this study is to determine whether BNC105P in combination with/following everolimus is effective in the treatment of progressive metastatic clear cell renal cell carcinoma following prior tyrosine kinase inhibitors.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Phase I: Patients will be accrued in the classic 3 patients per dose per cohort design, 21-day cycle

* Dose Level 1 Everolimus 10 mg BNC105P 4.2 mg/m2
* Dose Level 2 Everolimus 10 mg BNC105P 8.4 mg/m2
* Dose Level 3 Everolimus 10 mg BNC105P 12.6 mg/m2
* Dose Level 4 Everolimus 10 mg BNC105P 16 mg/m2

Phase II: Patients will be randomized 1:1 to Arm A or Arm B

Combination Arm A: Everolimus 10 mg + BNC105P MTD (from Phase 1 study) 21 day cycle

Sequential Arm B: Everolimus 10 mg 21 day cycle

* Patients to receive BNC105P monotherapy at 16 mg/m2 following progression or intolerable toxicity on everolimus therapy.

Karnofsky Performance Score (KPS) ≥70 within 7 days prior to registration for protocol therapy.

Life Expectancy: Not specified

Hematopoietic:

* White blood cell count (WBC) > 3.5 K/mm3
* Hemoglobin (Hgb) > 8.5 g/dL
* Platelets > 100 K/mm3
* Absolute neutrophil count (ANC) > 1.5 K/mm3

Hepatic:

* Total Bilirubin < 1.25 x ULN
* Aminotransferase (AST and ALT) < 2.5 x ULN

Renal:

* Serum Creatinine < 2.5 x ULN (upper limit normal)

Cardiovascular:

* No significant cardiovascular events within 6 months (CVA, CAD, peripheral arterial obstruction, arrhythmias, cardiac dysfunction) of registration for protocol therapy
* No history of clinical CHF or LVEF <50% by Echo (or MUGA) within 30 days prior to registration for protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of component (any percent) of clear cell RCC (renal cell carcinoma).
* Metastatic or locally advanced unresectable RCC. NOTE: Prior nephrectomy is not mandatory.
* Progressive disease after 1-2 prior VEGF-directed tyrosine kinase inhibitors (TKIs).
* Measurable disease according to RECIST and obtained by imaging within 30 days prior to registration for protocol therapy.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 4 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to registration for protocol therapy.

Exclusion Criteria:

* No active brain metastases. Patients with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis within 30 days prior to registration on protocol therapy. NOTE: A patient with prior brain metastasis are eligible if they have completed their radiation treatment for brain metastasis ≥30 days prior to registration for protocol therapy, are off steroids, and are asymptomatic.
* No other currently active malignancy.
* No treatment with any investigational agent within 14 days prior to registration for protocol therapy. NOTE: If treated with investigational agent within 14 days prior to registration, AE must be resolved back to baseline.
* Prior cancer treatment must be completed at least 14 days prior to registration for protocol therapy and the patient must have recovered from the acute toxic effects of the regimen. With the exception of Bevacizumab treatment, which must be completed 30 days prior to registration for protocol therapy.
* Prior radiation therapy to < 25% of the bone marrow [see bone marrow radiation chart in the study procedure manual (SPM)] allowed if completed within 30 days prior to registration for protocol therapy.
* Corrected QT interval (QTc) ≤ 450 msec at least 7 days prior to registration for protocol therapy.
* No clinically significant infections as judged by the treating investigator.
* No liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
* No collecting duct, medullary or sarcomatoid histology.
* No prior treatment with temsirolimus or everolimus in the phase II component of the study. NOTE: Prior treatment with these agents is permitted in the phase I component of the study.
* No use of full dose, therapeutic anti-coagulation with warfarin or related anti-coagulants or unfractionated or low molecular weight heparins.
* No uncontrolled hypertension (BP >150/100mmHg despite full doses of 1 anti-hypertensive medication).
* No thrombotic event within 6 months (deep vein thrombosis, pulmonary embolism) of registration for protocol therapy.
* No grade 2 or greater peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hutson, D.O., Study Chair — Hoosier Cancer Research Network
Locations (108):
- United States (94):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Providence Health System: Roy and Patricia Disney Family Cancer Center, Burbank, California
  - Compassionate Cancer Care Medical Group, Inc., Corona, California
  - Compassionate Cancer Care Medical Group, Corona, California
  - City of Hope, Duarte, California
  - Robert A. Moss, M.D., FACP, Inc., Fountain Valley, California
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Marin Specialty Care, Greenbrae, California
  - Good Samaritan Hospital, Los Angeles, California
  - UCLA Med - Hematology & Oncology, Los Angeles, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - American Institute of Research, Whittier, California
  - Centura Health Research Center, Denver, Colorado
  - Western Oncology & Hematology, Golden, Colorado
  - Cancer Care Centers of Florida: Brooksville, Brooksville, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - University of Florida, Shands Cancer Center, Gainesville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Cancer Care Centers of Florida, New Port Richey, Florida
  - Ocala Cancer Institute, Ocala, Florida
  - Cancer Care Centers of Brevard, Rockledge, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Dublin Hematology & Oncology Care, Dublin, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Edward H. Kaplan, M.D., & Associates, Skokie, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - IU Health Goshen, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Research, Lafayette, Indiana
  - IU Health at Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Oncology Hematology Associates of SW Indiana, Newburgh, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Siouxland Hematology Oncology Associates, LLP, Nylen Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Purchase Cancer Group, Paducah, Kentucky
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Metairie Oncologists, Metairie, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Metro Health Cancer Care, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Bozeman Deaconness Cancer Center, Bozeman, Montana
  - Sletten Cancer Specialists, Great Falls, Montana
  - Methodist Cancer Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Manchester, New Hampshire
  - Trinitas Regional Medical Center, Elizabeth, New Jersey
  - Somerset Hematology Oncology Associates, Somerville, New Jersey
  - Presbyterian Medical Group, Albuquerque, New Mexico
  - University of New Mexico Cancer Center: Albuquerque, Albuquerque, New Mexico
  - New York Oncology Hematology, PC, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Arena Oncology, Lake Success, New York
  - Tisch Cancer Institute at Mount Sinai Medical Center, New York, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - First Health of the Carolinas, Pinehurst, North Carolina
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Lawrence M. Stallings, M.D., Wooster, Ohio
  - Mercy Physicians Of Oklahoma, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute, Springfield, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Berks Hematology Oncology Associates, West Reading, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island, Cranston, Rhode Island
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - The Jones Clinic, PC, Germantown, Tennessee
  - Texas Oncology: Austin North, Austin, Texas
  - Texas Oncology: Bedford, Bedford, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Texas Oncology: Fort Worth, Fort Worth, Texas
  - Texas Oncology: Houston Memorial City, Houston, Texas
  - Methodist Hospital Research Institute, Houston, Texas
  - Houston Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - CTRC at The UT Health Science Center at San Antonio, San Antonio, Texas
  - Lynchburg Hematology Oncology Clinic, Inc., Lynchburg, Virginia
  - Harrison HealthPartners Bremerton Hematology & Oncology, Bremerton, Washington
  - Cascade Cancer Center, Kirkland, Washington
  - Group Health Medical Centers, Seattle, Washington
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington
  - Rockwood Clinic, Spokane, Washington
  - University of Wisconsin, Clinical Cancer Center, Milwaukee, Wisconsin
- Australia (13):
  - Royal Prince Alfred Hospital: Sydney Cancer Centre, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Sydney Adventist Hospital Ltd., Wahroonga, New South Wales
  - Gallipoli Medical Research Foundation: Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ashford Cancer Centre, Kurralta Park, South Australia
  - Gallipoli Medical Research Foundation: Launceston General Hospital, Launceston, Tasmania
  - Peninsula Oncology Centre, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- National Cancer Centre Singapore, Singapore, Singapore

REFERENCES:
- [Result] Thomas E. Hutson, Long H. Dang, Richard C. Lauer, Alexander Starodub, Ralph J. Hauke, Matt D. Galsky, Kathryn A. Bylow, Theodore Logan, Charles Lance Cowey, David C. Bibby, Gabriel Kremmidiotis, Elizabeth E. Doolin, Tina C. Lavranos, Guru Sonpavde, Noah M. Hahn, Christopher Sweeney, John Sarantopoulos. Phase I results of a phase I/II trial of BNC105P with everolimus in metastatic renal cell carcinoma (mRCC) patients previously treated with VEGFR tyrosine kinase inhibitors. J Clin Oncol 30, 2012 (suppl; abstr 4603) http://www.asco.org/ASCOv2/Meetings/Abstracts&vmview=abst_detail_view&confID=114&abstractID=91911
- [Result] John Sarantopoulos, Long H. Dang, Richard C. Lauer, Alexander Starodub, Ralph J. Hauke, Matt D. Galsky, Kathryn A. Bylow, Charles Lance Cowey, David C. Bibby, Gabriel Kremmidiotis, Elizabeth E. Doolin, Tina C. Lavranos, Jose Luis Iglesias, Guru Sonpavde, Theodore Logan, Noah M. Hahn, Christopher Sweeney, Thomas E. Hutson. A phase I/II trial of BNC105P with everolimus in metastatic renal cell carcinoma (mRCC) patients: Updated phase I results of the Disruptor-1 trial. J Clin Oncol 31, 2013 (suppl; abstr 4563. http://abstracts2.asco.org/AbstView_132_107981.html
- [Result] Pal S, Azad A, Bhatia S, Drabkin H, Costello B, Sarantopoulos J, Kanesvaran R, Lauer R, Starodub A, Hauke R, Sweeney CJ, Hahn NM, Sonpavde G, Richey S, Breen T, Kremmidiotis G, Leske A, Doolin E, Bibby DC, Simpson J, Iglesias J, Hutson T. A Phase I/II Trial of BNC105P with Everolimus in Metastatic Renal Cell Carcinoma. Clin Cancer Res. 2015 Aug 1;21(15):3420-7. doi: 10.1158/1078-0432.CCR-14-3370. Epub 2015 Mar 18. PMID 25788492
- [Derived] Yang ES, Nassar AH, Adib E, Jegede OA, Alaiwi SA, Manna DLD, Braun DA, Zarei M, Du H, Pal SK, Naik G, Sonpavde GP. Gene Expression Signature Correlates with Outcomes in Metastatic Renal Cell Carcinoma Patients Treated with Everolimus Alone or with a Vascular Disrupting Agent. Mol Cancer Ther. 2021 Aug;20(8):1454-1461. doi: 10.1158/1535-7163.MCT-20-1091. Epub 2021 Jun 9. PMID 34108261
- See also: Hoosier Cancer Research Network Homepage — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Participants: Participants in the phase I dose escalation portion of the study.
- Phase II: Arm A: Phase II Participants, Arm A
  Everolimus 10mg + BNC105P(Phase I MTD)
- Phase II: Arm B Participants: Phase II: Arm B Participants
  Everolimus 10mg followed by BNC105P monotherapy (16mg/m^2) following progression or intolerable toxicity on Everolimus therapy.
Period: Phase I
Arm/Group | Phase I Participants | Phase II: Arm A | Phase II: Arm B Participants
Started | 15 | 0 (No Phase II Participants were enrolled during this time period) | 0 (No Phase II Participants were enrolled during this time period)
Completed | 12 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Symptomatic Deterioration before Treatme | 3 | 0 | 0
Period: Phase II
Arm/Group | Phase I Participants | Phase II: Arm A | Phase II: Arm B Participants
Started | 0 (No Phase I Participants were enrolled during this time period.) | 70 | 69
Completed | 0 | 69 | 67
Not Completed | 0 | 1 | 2
Not completed — Not Evaluable per protocol | 0 | 0 | 2
Not completed — Determined Ineligible per protocol | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II: Arm A: Phase II Participants, Arm A
  Everolimus + BNC105P
- Phase II: Arm B Participants: Phase II: Arm B Participants
  Everolimus only, followed by BNC105P monotherapy
- Total: Total of all reporting groups
Arm/Group | Phase I Participants | Phase II: Arm A | Phase II: Arm B Participants | Total
Number analyzed (Participants) | 15 | 69 | 69 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9) | 62 (9) | 63 (9) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 20 | 13 | 39
  Male | 9 | 49 | 56 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 8
  White | 13 | 61 | 59 | 133
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Initial Karnovksy Performance Score (KPS) [Count of Participants; unit: Participants] — Karnofsky Performance Status (KPS) is a general indicator of a subject's well being and ability to carry on daily activities. The KPS scale ranges from 0-100 in 10 unit increments where 100=Normal; no complaints; no evidence of disease and 0=Dead
  Participants
    KPS 100 | 0 | 29 | 25 | 54
    KPS 90 | 9 | 23 | 24 | 56
    KPS 80 | 2 | 13 | 15 | 30
    KPS 70 | 4 | 4 | 5 | 13
Memorial Sloan Kettering Cancer Center Risk Group (MSKCC [Count of Participants; unit: Participants]
  MSKCC Risk Group - Good | 3 | 17 | 16 | 36
  MSKCC Risk Group - Intermediate | 11 | 45 | 47 | 103
  MSKCC Risk Group - Poor | 1 | 7 | 6 | 14
Metastatic Site [Count of Participants; unit: Participants]
  Lung | 13 | 57 | 54 | 124
  Liver | 6 | 13 | 13 | 32
  Bone | 8 | 21 | 24 | 53
  Brain | 2 | 3 | 5 | 10
Number of Prior Therapies [Count of Participants; unit: Participants]
  1 Prior Therapy | 0 | 14 | 13 | 27
  2 Prior Therapies | 0 | 24 | 18 | 42
  3 Prior Therapies | 3 | 10 | 15 | 28
  >=4 Prior Therapies | 12 | 21 | 23 | 56

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose of BNC105P in Combination With Everolimus.
Description: Phase I
Time Frame: Until disease progression or unacceptable toxicity, up to 24 cycles or 24 months
Population: 12 participants completed at least one cycle of combination therapy and were evaluable.
Measure: Number; unit: mg/m^2
Groups:
- Phase I Participants: 15 total Participants were recruited to the phase I portion of the study.
Arm/Group | Phase I Participants
Number analyzed (Participants) | 12
mg/m^2 | 16

2. Primary Outcome: Phase I: Toxicities of BNC105P in Combination With Everolimus.
Description: Determine the toxicities of BNC105P in combination with everolimus. Drug-related treatment emergent adverse events by CTCAE grade 2 or greater are reported
Time Frame: Until disease progression or unacceptable toxicity, up to 24 cycles or 24 months
Population: 12 participants who completed at least one cycle of combination therapy.
Measure: Number; unit: participants
Arm/Group | Phase I Participants
Number analyzed (Participants) | 12
participants
  AST-SGOT Grade 2 | 1
  Cough Grade 2 | 1
  Dyspepsia Grade 2 | 1
  Hemoglobin Grade 2 | 4
  Hemoglobin Grade 3 | 1
  Hypomagnesia Grade 2 | 1
  Low Platelets Grade 2 | 1
  Weight Loss Grade 2 | 1
  Fatigue Grade 2 | 2
  Left ventricular systolic dysfunction Grade 2 | 1
  Mucositis (oral) Grade 2 | 2
  Nail Infection Grade 2 | 1
  Diaphoresis Grade 2 | 1
  Pericardial effusion Grade 3 | 1
  Pleural effusion Grade 2 | 1

3. Primary Outcome: Phase II: 6-month Progression Free Survival (PFS) With the Addition of BNC105P to Everolimus.
Description: Improvement in 6-month PFS with the addition of BNC105P to everolimus. Progression is defined using RECIST criteria as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 6 months
Measure: Number; unit: probability of 6MPFS
Groups:
- Sequential Arm B:Everolimus Followed by BNC105P Monotherapy: Sequential Arm B: Everolimus 10 mg, 21 day cycle
  Patients to receive BNC105P monotherapy at 16 mg/m2 following progression or intolerable toxicity on everolimus therapy.
  Everolimus: Everolimus 10 mg. Taken orally, every evening, 1 hr before or 2 hrs after meals
  BNC105P: BNC105P, up to 16 mg/m^2
Arm/Group | Combination Arm A: Everolimus + BNC105P | Sequential Arm B:Everolimus Followed by BNC105P Monotherapy
Number analyzed (Participants) | 69 | 67
probability of 6MPFS | .3382 | .3030
Statistical Analysis 1: Comparison: Combination Arm A: Everolimus + BNC105P vs Sequential Arm B:Everolimus Followed by BNC105P Monotherapy; Test type: Other; p = .6625, Chi-squared

4. Secondary Outcome: Phase I: Response Rate of BNC105P in Combination With Everolimus.
Description: Number of objective responses per RECIST criteria. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Until disease progression or unacceptable toxicity, up to 24 cycles or 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Participants
Number analyzed (Participants) | 15
Participants
  CR | 0
  PR | 0
  SD | 8
  PD | 4
  Unknown | 3

5. Secondary Outcome: Geometric Mean Half-life of BNC105 and BNC105P in Combination With Everolimus.
Description: Determine the PK Profile for BN105P in combination with everolimus by calculating the geometric mean half-life of BNC105P
Time Frame: 12 months
Population: 14 participants has sufficient data collected for the analysis of this objective
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Phase I Participants
Number analyzed (Participants) | 14
hours
  Half-life of BNC105 | .32 [.16 to 1.65]
  Half-life of BNC105P | .08 [.05 to .13]

6. Secondary Outcome: Phase II: Response Rate With Combination Therapy Compared to Everolimus Alone
Description: Objective response is defined as a confirmed CR or PR per RECIST criteria. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Arm A: Everolimus + BNC105P | Sequential Arm B:Everolimus Followed by BNC105P Monotherapy
Number analyzed (Participants) | 69 | 67
Participants | 1 | 1

7. Secondary Outcome: Phase II: Progression Free Survival (PFS) With BNC105P Alone in Patients After Progressing on Everolimus.
Description: Median time to progression for arm P participants who crossed over to BNC105P monotherapy after progression. Progression is defined per RECIST criteria as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm B Participants Who Crossed Over to BNC105P Monotherapy: After progression on everolimus, 33 participants crossed over to BNC105P monotherapy per protocol.
Arm/Group | Arm B Participants Who Crossed Over to BNC105P Monotherapy
Number analyzed (Participants) | 25
months | 1.8 [1.74 to 2.04]

8. Secondary Outcome: Phase II: Adverse Events of Everolimus and BNC105P When Administered as a Combination or Sequential Regimen.
Description: Determine adverse events of everolimus and BNC105P when administered as a combination or sequential regimen. Total number of serious and non-serious adverse events for Arm A and Arm B are summarized. Complete adverse event information is supplied in the Adverse Events reporting section.
Time Frame: 12 months
Measure: Number; unit: number of adverse events
Arm/Group | Combination Arm A: Everolimus + BNC105P | Sequential Arm B:Everolimus Followed by BNC105P Monotherapy
Number analyzed (Participants) | 69 | 67
number of adverse events
  Non-Serious Adverse Events | 1419 | 1654
  Serious Adverse Events | 39 | 50

9. Secondary Outcome: Phase II: Overall Survival
Description: Determine overall survival probability, up to a maximum of 5 years from registration for protocol therapy.
Time Frame: 60 months
Measure: Number; unit: probability of OS at 60 months.
Arm/Group | Combination Arm A: Everolimus + BNC105P | Sequential Arm B:Everolimus Followed by BNC105P Monotherapy
Number analyzed (Participants) | 69 | 67
probability of OS at 60 months. | .15 | .21

10. Secondary Outcome: Exploratory Objective: Correlation of PFS With Biomarkers
Description: Exploratory analysis of serum biomarkers were undertaken to generate a potential signature for response. The correlation with 6 month progression free survival P value for four plasma biomarkers is reported.
Time Frame: 6 months
Population: Analysis was pre-specified to look at the correlation irrespective of arm.
Measure: Number; unit: Correlation with PFS P Value
Groups:
- Phase II Participants With Sufficient Correlative Samples: A subset of Phase II Participants who had sufficient correlative samples drawn for plasma biomarker analysis.
Arm/Group | Phase II Participants With Sufficient Correlative Samples
Number analyzed (Participants) | 44
Correlation with PFS P Value
  Serum Amyloid P-Component (SAP) | 0.0184
  Sex Hormone-Binding Globulin (SHBG) | 0.0063
  Matrix Metalloproteinase-9 (MMP-9) | 0.0421
  Stem Cell Factor (SCF) | 0.0291

ADVERSE EVENTS:
Time Frame: 60 Months
Groups:
- Phase II: Arm A: Phase II Participants, Arm A
- Phase II: Arm B Participants: Phase II: Arm B Participants
Arm/Group | Phase I Participants | Phase II: Arm A | Phase II: Arm B Participants
Serious Adverse Events (participants affected / at risk) | 9/15 | 22/70 | 31/69
Other Adverse Events (participants affected / at risk) | 15/15 | 70/70 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Participants (N=15) | Phase II: Arm A (N=70) | Phase II: Arm B Participants (N=69)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Investigations) | 1 (1) | 0 (0) | 2 (3)
CARDIAC GENERAL (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
DEATH NOT ASSOCIATED WITH CTCAE TERM / MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 0 (0) | 0 (0) | 2 (2)
FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 0 (0) | 1 (1) | 1 (1)
HEMOGLOBIN (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
HEMORRHAGE, GU / URINARY NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / RECTUM (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC / LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
LYMPHATICS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
OBSTRUCTION, GI / SMALL BOWEL NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN / BACK (General disorders) | 0 (0) | 2 (2) | 1 (1)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN / NECK (General disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN / TUMOR PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL ARTERIAL ISCHEMIA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 0 (0) | 1 (1) | 0 (0)
PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 3 (4)
RENAL FAILURE (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)
RENAL/GENITOURINARY (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 0 (0) | 0 (0) | 2 (2)
THROMBOSIS/EMBOLISM (VASCULAR ACCESS-RELATED) (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VASCULAR (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Participants (N=15) | Phase II: Arm A (N=70) | Phase II: Arm B Participants (N=69)
ACIDOSIS (METABOLIC OR RESPIRATORY) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 2 (3) | 7 (11) | 7 (8)
ALKALINE PHOSPHATASE (Investigations) | 5 (6) | 10 (14) | 14 (19)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 (3) | 2 (5) | 2 (2)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 4 (4) | 4 (4) | 7 (7)
ALLERGY/IMMUNOLOGY (Immune system disorders) | 4 (5) | 0 (0) | 5 (6)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (2) | 8 (14) | 8 (13)
ANOREXIA (Gastrointestinal disorders) | 4 (7) | 16 (18) | 18 (21)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (14) | 5 (5)
ASCITES (NON-MALIGNANT) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 2 (6) | 9 (18) | 9 (12)
ATAXIA (INCOORDINATION) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
AUDITORY/EAR (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2)
AUTOIMMUNE REACTION (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
BICARBONATE, SERUM-LOW (Investigations) | 1 (2) | 0 (0) | 2 (3)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (1) | 0 (0) | 1 (2)
BLOOD/BONE MARROW (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 4 (4)
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 2 (2)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Investigations) | 2 (6) | 4 (4) | 7 (18)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (1) | 8 (12) | 6 (7)
CARDIAC ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
CARDIAC GENERAL (Cardiac disorders) | 1 (1) | 3 (6) | 4 (7)
CATARACT (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
CERVICAL SPINE-RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CHELITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 8 (9) | 22 (39) | 30 (40)
COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CONFUSION (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 6 (9) | 15 (17) | 27 (33)
CONSTITUTIONAL SYMPTOMS (General disorders) | 2 (5) | 3 (3) | 6 (11)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 28 (35) | 25 (36)
CREATININE (Investigations) | 5 (7) | 15 (26) | 13 (24)
CYSTITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 2 (2) | 2 (3) | 3 (3)
DENTAL: TEETH (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 1 (3) | 13 (17) | 16 (45)
DIARRHEA (Gastrointestinal disorders) | 7 (8) | 24 (37) | 17 (21)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (2) | 3 (3) | 6 (6)
DRY EYE SYNDROME (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 3 (3) | 2 (2) | 7 (7)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 7 (7)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (3)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 26 (32) | 27 (37)
EDEMA: HEAD AND NECK (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
EDEMA: LIMB (Blood and lymphatic system disorders) | 4 (4) | 18 (33) | 16 (22)
EDEMA: TRUNK/GENITAL (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ENDOCRINE (Endocrine disorders) | 1 (1) | 2 (3) | 3 (4)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 4 (4)
ESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (3) | 3 (3)
EXTRAPYRAMIDAL/INVOLUNTARY MOVEMENT/RESTLESSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 12 (27) | 42 (60) | 46 (83)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 5 (11) | 9 (11) | 13 (17)
FIBROSIS-DEEP CONNECTIVE TISSUE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
FLUSHING (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 1 (1) | 4 (5) | 4 (5)
GASTROINTESTINAL (Gastrointestinal disorders) | 3 (7) | 7 (11) | 9 (12)
GGT (GAMMA-GLUTAMYL TRANSPEPTIDASE) (Investigations) | 0 (0) | 2 (8) | 4 (9)
GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 3 (3) | 19 (51) | 24 (62)
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Investigations) | 0 (0) | 3 (6) | 2 (2)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
HEARING: PATIENTS WITHOUT BASELINE AUDIOGRAM AND NOT ENROLLED IN A MONITORING PROGRAM (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 4 (6) | 5 (5) | 15 (16)
HEMOGLOBIN (Blood and lymphatic system disorders) | 11 (49) | 35 (107) | 38 (99)
HEMOGLOBINURIA (Investigations) | 0 (0) | 1 (1) | 1 (1)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 2 (6)
HEMORRHAGE, GI / RECTUM (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HEMORRHAGE, GU / URINARY NOS (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (2)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / BRONCHOPULMONARY NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / LUNG (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7) | 9 (13)
HEMORRHAGE/BLEEDING (General disorders) | 0 (0) | 1 (1) | 3 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HOT FLASHES/FLUSHES (Endocrine disorders) | 1 (1) | 2 (2) | 1 (2)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 0 (0)
HYPERTENSION (Cardiac disorders) | 9 (9) | 23 (26) | 25 (27)
HYPOTENSION (Cardiac disorders) | 0 (0) | 2 (3) | 3 (3)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (2)
ILEUS, GI (FUNCTIONAL OBSTRUCTION OF BOWEL, I.E., NEUROCONSTIPATION) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INCONTINENCE, ANAL (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
INCONTINENCE, URINARY (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / BLADDER (URINARY) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTIONWITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / SINUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / SKIN (CELLULITES) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
INFECTIONWITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / URINARY TRACT NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 2 (3) | 5 (6) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / ABDOMEN NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BRONCHUS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / EXTERNAL EAR (OTITIS EXTERNA) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / EYE NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LARYNX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 2 (4) | 2 (3)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / ORAL CAVITY-GUMS (GINGIVITIS) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SINUS (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (3) | 1 (1) | 3 (3)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UNGUAL (NAILS) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UPPER AIRWAY NOS (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 1 (2) | 3 (4) | 1 (1)
INFECTION WITH UNKNOWN ANC / SINUS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC / SKIN (CELLULITES) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
INFECTION WITH UNKNOWN ANC / UPPER AIRWAY NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION WITH UNKNOWN ANC / URINARY TRACT NOS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
INFECTION WITH UNKNOWN ANC / VAGINA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INR (INTERNATIONAL NORMALIZED RATIO OF PROTHROMBIN TIME) (Surgical and medical procedures) | 0 (0) | 2 (3) | 1 (1)
INSOMNIA (General disorders) | 2 (2) | 14 (18) | 17 (18)
JOINT-FUNCTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 3 (4) | 4 (16) | 5 (15)
LIPASE (Investigations) | 0 (0) | 0 (0) | 1 (1)
LIVER DYSFUNCTION/FAILURE (CLINICAL) (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
LUMBAR SPINE-RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
LYMPHATICS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (4)
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 (7) | 5 (13) | 4 (8)
MAGNESIUM, SERUM-HIGH (HYPERMAGNESEMIA) (Investigations) | 1 (1) | 0 (0) | 1 (1)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 1 (1) | 2 (2) | 4 (4)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
METABOLIC/LABORATORY (Investigations) | 3 (3) | 9 (22) | 11 (24)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 2 (3) | 5 (5) | 8 (9)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 1 (1) | 6 (6) | 9 (9)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 3 (3) | 13 (20) | 21 (41)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / PHARYNX (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / STOMACH (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 1 (1) | 11 (11) | 9 (28)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTRAOCULAR (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 3 (3)
MUSCULOSKELETAL/SOFT TISSUE (Musculoskeletal and connective tissue disorders) | 7 (15) | 8 (11) | 13 (20)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3) | 2 (3)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 9 (11) | 18 (20) | 21 (27)
NEUROENDOCRINE: ADH SECRETION ABNORMALITY (E.G., SIADH OR LOW ADH) (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
NEUROLOGY (Nervous system disorders) | 1 (1) | 1 (1) | 2 (5)
NEUROPATHY: MOTOR (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
NEUROPATHY: SENSORY (Nervous system disorders) | 0 (0) | 6 (6) | 3 (4)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 7 (15) | 8 (16)
OBESITY (General disorders) | 0 (0) | 1 (1) | 0 (0)
OCULAR SURFACE DISEASE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
OCULAR/VISUAL (Eye disorders) | 4 (5) | 3 (4) | 2 (5)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 4 (4) | 11 (12) | 10 (15)
PAIN / ANUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN / BACK (General disorders) | 6 (11) | 15 (18) | 22 (35)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 2 (7) | 5 (7) | 9 (15)
PAIN / BREAST (Reproductive system and breast disorders) | 1 (4) | 1 (1) | 0 (0)
PAIN / BUTTOCK (General disorders) | 0 (0) | 1 (1) | 3 (3)
PAIN / CARDIAC/HEART (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (10) | 11 (22)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 6 (7) | 7 (9)
PAIN / EXTERNAL EAR (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 2 (2)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 4 (7) | 17 (26) | 13 (18)
PAIN / EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN / FACE (General disorders) | 0 (0) | 2 (3) | 1 (2)
PAIN / HEAD/HEADACHE (General disorders) | 3 (4) | 7 (8) | 17 (22)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 3 (4) | 9 (9) | 6 (7)
PAIN / KIDNEY (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
PAIN / LIP (General disorders) | 0 (0) | 2 (2) | 0 (0)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 3 (3)
PAIN / NECK (General disorders) | 0 (0) | 3 (4) | 2 (2)
PAIN / ORAL CAVITY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
PAIN / ORAL-GUMS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
PAIN / PAIN NOS (General disorders) | 0 (0) | 0 (0) | 1 (3)
PAIN / PELVIS (General disorders) | 0 (0) | 0 (0) | 2 (2)
PAIN / PHANTOM (PAIN ASSOCIATED WITH MISSING LIMB) (General disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN / SCALP (General disorders) | 0 (0) | 1 (1) | 1 (1)
PAIN / STOMACH (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 4 (4)
PAIN / TUMOR PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN / URETHRA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 7 (12) | 10 (18) | 9 (16)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC ENDOCRINE: GLUCOSE INTOLERANCE (Endocrine disorders) | 2 (2) | 2 (3) | 2 (2)
PERICARDIAL EFFUSION (NON-MALIGNANT) (Cardiac disorders) | 4 (6) | 0 (0) | 1 (1)
PERSONALITY/BEHAVIORAL (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
PHOSPHATE, SERUM-LOW (HYPOPHOSPHATEMIA) (Investigations) | 3 (4) | 6 (6) | 7 (10)
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PLATELETS (Blood and lymphatic system disorders) | 7 (12) | 23 (36) | 11 (16)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 3 (5) | 3 (3)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (5) | 3 (6)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 2 (3) | 4 (4) | 4 (10)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 2 (5) | 9 (21) | 5 (6)
PROTEINURIA (Investigations) | 4 (15) | 11 (17) | 12 (16)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 3 (4) | 11 (12) | 5 (12)
PSYCHOSIS (HALLUCINATIONS/DELUSIONS) (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PTT (PARTIAL THROMBOPLASTIN TIME) (Surgical and medical procedures) | 1 (1) | 3 (3) | 0 (0)
PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8) | 7 (24)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (2) | 15 (19) | 16 (21)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2) | 11 (14) | 8 (10)
RASH: DERMATITIS ASSOCIATED WITH RADIATION / RADIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 4 (8)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
RENAL/GENITOURINARY (Renal and urinary disorders) | 3 (3) | 15 (21) | 14 (17)
RIGORS/CHILLS (General disorders) | 3 (3) | 3 (5) | 6 (8)
SALIVARY GLAND CHANGES/SALIVA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
SEROMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SODIUM, SERUM-HIGH (HYPERNATREMIA) (Investigations) | 1 (1) | 1 (2) | 2 (3)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 5 (10) | 10 (15) | 12 (16)
STRICTURE/STENOSIS (INCLUDING ANASTOMOTIC), GU / PROSTATE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
SWEATING (DIAPHORESIS) (General disorders) | 3 (5) | 5 (6) | 5 (5)
SYNDROMES (General disorders) | 0 (0) | 1 (1) | 0 (0)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 3 (3) | 5 (8) | 11 (12)
THROMBOSIS/EMBOLISM (VASCULAR ACCESS-RELATED) (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
THYROID FUNCTION, HIGH (HYPERTHYROIDISM, THYROTOXICOSIS) (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
THYROID FUNCTION, LOW (HYPOTHYROIDISM) (Endocrine disorders) | 3 (3) | 3 (3) | 9 (9)
TRIGLYCERIDE, SERUM-HIGH (HYPERTRIGLYCERIDEMIA) (Investigations) | 6 (6) | 21 (54) | 28 (74)
ULCER, GI / DUODENUM (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (3)
URIC ACID, SERUM-HIGH (HYPERURICEMIA) (Investigations) | 0 (0) | 0 (0) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 0 (0) | 2 (2) | 5 (5)
URINE COLOR CHANGE (Renal and urinary disorders) | 1 (1) | 2 (3) | 0 (0)
URTICARIA (HIVES, WELTS, WHEALS) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
VAGINITIS (NOT DUE TO INFECTION) (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
VASCULAR (Vascular disorders) | 1 (2) | 0 (0) | 1 (1)
VESSEL INJURY-VEIN / SVC (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 2 (2) | 3 (3) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
VOMITING (Gastrointestinal disorders) | 5 (5) | 8 (8) | 13 (16)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
WEIGHT LOSS (General disorders) | 7 (8) | 5 (6) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No